CLINICAL TRIAL: NCT05515380
Title: Performance Evaluation of the Tennis Serve Using 8-stage Model and Its Implications in National Pakistani Tennis Players
Brief Title: 8-stage Model and Its Implications in National Pakistani Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/01024 Ali Zubair
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Sports Physical Therapy
Keywords: 8-Stage Model; Flexibility; Strength; Tennis Serve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-stage model based exercise training (Experimental): 8-stage model based exercise training
  Interventions: Other: 8-stage model based exercise program
- Conventional exercise training (Active Comparator): Conventional exercise training
  Interventions: Other: Conventional exercise program

INTERVENTIONS:
Other: 8-stage model based exercise program — The experimental group would follow exercises related to 8 phases of tennis serve, which would be based on 8-stage model. The participants would follow this program for three days per week for 12 weeks.
  Arms: 8-stage model based exercise training
Other: Conventional exercise program — The control group would follow conventional exercise program advised by coaches. The participants of this group would also follow this program for three days per week for 12 weeks.
  Arms: Conventional exercise training

SUMMARY:
The aim of this study is to determine the effectiveness of structured exercises for tennis serve performance by using 8-stage model.

DETAILED DESCRIPTION:
Tennis serve stroke is the most crucial component of tennis. 8-stage model like other training programs has proven to be effective in improving performance. This exercise program has yet not been implemented in Pakistani tennis players and remain to be tested in local population.

This randomized controlled trial has been designed to assess the effectiveness of 8-stage model based exercise program in Pakistani national tennis players. The present study has hypothesized that there will be a significant difference between the effects of 8-stage model and conventional training program. There are two arms of intervention in this study: experimental and control group. Experimental group would follow the 8-stage model based exercise training program while control group would follow their conventional exercise training program. Outcome measurements (speed, flexibility, strength) has been carried out at baseline and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* National level tennis players
* Players who are playing tennis from last one year continuously

Exclusion Criteria:

* Players with any MSK injury
* Any systemic disease affecting players performance
* Any inflammatory conditions.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Serve speed | Change from Baseline at 12th week
  Serve speed will be measured using Bushnell's Velocity Speed Gun. Speed gun is used to measure the speed of tennis ball in tennis court. It measures around 6-200 miles speed of ball with accuracy along with distance of ball as far as 90 feet away.
Upper limbs' flexibility | Change from Baseline at 12th week
  Shoulder flexibility will be measured based on recommendations by International Tennis Federation (ITF) and range of motion through Goniometer. The overall upper limb flexibility was measured using shoulder and wrist flexibility test recommended by ITF. The range of motion measurement would include combined range of motion of external and internal rotation.
Upper limbs' strength | Change from Baseline at 12th week
  Shoulder strength will be measured based on recommendations by International Tennis Federation (ITF) and wrist strength through hand held dynamometer. The overall upper limb strength was measured using shoulder push up test recommended by ITF. The wrist strength measurement would include maximum force produced using hand held wrist dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Noman Sadiq, MS-SPT, Principal Investigator — Riphah International University, Islamabad.
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No